CLINICAL TRIAL: NCT06044129
Title: A Novel Approach Integrating Magnetic Resonance Imaging (MRI) Data and Artificial Intelligence for Predicting the Success Rate of Vaginal Delivery in Pregnant Women
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2023-07-209
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaginal trial labor group
  Interventions: Device: Mri scan of fetal head and pelvis

INTERVENTIONS:
Device: Mri scan of fetal head and pelvis — The pelvic parameters and fetal head parameters of pregnant women were measured by MRI, including pelvic entrance plane, middle pelvic plane, pelvic outlet plane, pubic arch Angle, double parietal diameter, occipitofrontal diameter, and suboccipital fontanel diameter.

SUMMARY:
The aim of this study was to use MRI imaging to accurately scan the pregnant woman's pelvis and fetal skull, build a 3D model of them, and combine with artificial intelligence to develop an accurate tool to predict the success rate of vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Full-term.
* Single fetus, head first.
* Pregnant women have vaginal couvade wishes.
* Complete clinical data of pregnant women.

Exclusion Criteria:

* Pregnancy with serious medical and surgical diseases.
* Abnormal fetal position (such as transverse, breech, etc.).
* Twin or multiple pregnancies.
* Vaginal couvade contraindications such as placenta previa.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Full-term single live pregnant women who gave birth in the Department of Obstetrics of the Second Affiliated Hospital of Wenzhou Medical University from January 1, 2024 to December 31, 2026 were selected as the study population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The mode of delivery | during delivery
  Vaginal or cesarean delivery in the end

CONTACTS AND LOCATIONS:
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China